CLINICAL TRIAL: NCT06558721
Title: Comparison of the Effectiveness of Mirror Therapy and Functional Electrical Stimulation Bicycle Ergometry Therapy Applied to the Lower Extremity in Stroke Patients
Brief Title: Effectiveness of Functional Electric Stimulation With Bicycle Ergometer and Mirror Therapy in Stroke Patients Lower Extremity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Muhammed Sefa Cınar, Asist. Dr., Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1-23-4032
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: Stroke; Lower Extremity; Mirror Therapy; Functional Electric Stimulation; Bicycle Ergometer
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional Rehabilitation (Active Comparator): Lower extremity conventional rehabilitation in stroke patients
  Interventions: Other: Conventional rehabilitation
- Conventional Rehabilitation + Mirror Therapy (Active Comparator): Mirror therapy in addition to conventional rehabilitation of the lower extremity in stroke patients
  Interventions: Other: Conventional rehabilitation; Other: Mirror therapy
- Conventional Rehabilitation + Bicycle Ergometer with Functional Electric Stimulation (Active Comparator): Bicycle Ergometer with Functional Electric Stimulation Therapy in addition to conventional rehabilitation of the lower extremity in stroke patients
  Interventions: Other: Conventional rehabilitation; Device: Bicycle ergometer with functional electric stimulation

INTERVENTIONS:
Other: Conventional rehabilitation — Lower extremity conventional rehabilitation in stroke patients
Other: Mirror therapy — Mirror therapy of the lower extremity in stroke patients
  Arms: Conventional Rehabilitation + Mirror Therapy
Device: Bicycle ergometer with functional electric stimulation — Bicycle ergometer with functional electric stimulation therapy of the lower extremity in stroke patients
  Arms: Conventional Rehabilitation + Bicycle Ergometer with Functional Electric Stimulation

SUMMARY:
There are different methods in stroke rehabilitation. In addition to conventional techniques, functional electric stimulation with bicycle ergometer therapy and mirror therapy can be used. In this study, we will compare functional electric stimulation with bicycle ergometer therapy and mirror therapy in stroke patients.

DETAILED DESCRIPTION:
Aim of study is to compare functional electric stimulation with bicycle ergometer therapy and mirror therapy applied to lower extremity in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 age
* Unilateral stroke
* First time stroke
* Time after stroke less than 6 months
* Lower extremity Brunnstrom stage: 2-4
* Lower extremity spasticity Modified Ashworth Scale: less than 3
* Patient with sitting balance
* Mini Mental Test Score higher than 23
* Patients signed approval form

Exclusion Criteria:

* Bilateral stroke
* Neurological disease other than stroke
* Psychiatric disease
* Lower extremity orthopedic problem
* Visual or audience problem
* Neglect
* Severe aphasia
* Contraindications of electrical stimulation (cardiac implantation etc.)
* Severe comorbidity (cardiac failure etc.)
* Seizure
* Acute deep vein thromboembolism
* Local infection
* Botulinum toxin injection of lower extremity less than 3 month

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Lower Extremity Motor Subscale | Before treatment (0. week), finishing time of treatment (6.week)

SECONDARY OUTCOMES:
Brunnstrom Staging | Before treatment (0. week), finishing time of treatment (6.week)
Berg Balance Scale | Before treatment (0. week), finishing time of treatment (6.week)
Functional Independence Measure - Motor Score | Before treatment (0. week), finishing time of treatment (6.week)
Stroke Specific Quality of Life Scale | Before treatment (0. week), finishing time of treatment (6.week)
Functional Ambulation Scale | Before treatment (0. week), finishing time of treatment (6.week)

CONTACTS AND LOCATIONS:
Overall Officials: Engin Koyuncu, Prof. Dr., Principal Investigator — Gaziler Physical Therapy and Rehabilitation Training and Research Hospital
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Training and Research Hospital, Ankara, Çankaya, Turkey (Türkiye)